CLINICAL TRIAL: NCT02781896
Title: Direct Left Ventricular Rapid Pacing Via the Valve Delivery Guide-wire in TAVI: a Randomized Study
Brief Title: Direct Left Ventricular Rapid Pacing Via the Valve Delivery Guide-wire in TAVI
Acronym: EASY TAVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier Mutualiste de Grenoble (Other)
Collaborators: Centre Recherche Cardio Vasculaire Alpes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: EASY TAVI 2016
Record Dates: First submitted 2016-05-18; First posted 2016-05-25 (Estimated); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Aortic Valve Stenosis
Keywords: TAVI; aortic valve bioprothesis; TAVI simplification; aortic stenosis; rapid left ventricular pacing; TAVR
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Right ventricular pacing (Active Comparator): Rapid pacing during TAVI is provided by a temporary pacing catheter placed in the right ventricle. An additional venous vascular access is required.
  Interventions: Device: pacing catheter
- Left ventricular pacing (Experimental): Rapid pacing during TAVI is provided by the valve delivery guidewire inserted into the left ventricle using two alligator clamps. One clamp is attached directly to the skin at the femoral entry site, the other is attached to the body of the valve delivery guidewire. No additional venous vascular access is required.
  Interventions: Device: valve delivery guidewire

INTERVENTIONS:
Device: pacing catheter — Rapid pacing during TAVI is required to ensure transient cardiac standstill while predilatation is performed and the valve is being positioned and deployed. In the right ventricular pacing arm, rapid pacing is provided by a standard right ventricular pacing catheter.
  Other Names: transvenous stimulation electrode; pacing lead; pacing wire
  Arms: Right ventricular pacing
Device: valve delivery guidewire — Rapid pacing during TAVI is required to ensure transient cardiac standstill while predilatation is performed and the valve is being positioned and deployed. In the Left ventricular pacing arm, rapid pacing is provided via the valve-delivery guidewire inserted into the left ventricle. The cathode of an external pacemaker is placed on the external end of the guidewire using an alligator clamp. The TAVI catheter provides the necessary insulation. The anode is attached directly to the subcutaneous tissue at the femoral entry site (also using an alligator clamp).
  Arms: Left ventricular pacing

SUMMARY:
The purpose of this study is to determine whether a left ventricular rapid pacing using the valve delivery guide-wire in transcatheter aortic valve implantation (TAVI) reduces the overall procedure duration in comparison with the conventional method.

DETAILED DESCRIPTION:
Use of temporary pacing via a right ventricular lead in TAVI is still mandatory to ensure transient cardiac standstill while predilatation is performed and the valve is being positioned and deployed. This requires an additional venous vascular access and a pacing catheter which are both likely to generate complications.

This study compares the standard right ventricular rapid pacing to a new and simplified technique : a left ventricular rapid pacing is provided via the back-up 0.035 " guidewire. The cathode of an external pacemaker is placed on the tip of the 0.035" wire and the anode on a needle inserted into the groin. Insulation is ensured by the balloon or TAVI catheter.

ELIGIBILITY:
Inclusion Criteria:

* Subject is eligible for a TAVI
* Access considered for aortic valve bioprothesis delivery is transfemoral
* Aortic valve bioprothesis considered is Edwards Sapien 3® et/ou XT®
* Subject is ≥ 18 years of age
* Subject has signed informed consent form

Exclusion Criteria:

* Pregnancy
* Subject already included in this study
* Subject included in another study and whose inclusion in EASY TAVI implies a deviation in either study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-06-29 (Actual)

PRIMARY OUTCOMES:
Total TAVI procedural duration | 1 month
  Duration of TAVI procedure is calculated from the first puncture to the last sheath removal

SECONDARY OUTCOMES:
Efficacy of the experimental technique to create a blood pressure drop reaching at least 60 mmHg (Ventricular stimulation efficiency) | 1 month
  Stimulation efficiency is defined as a drop in systolic blood pressure reaching at least 60 mmHg during the prolonged stimulation without loss of capture for more than 30s.
Incidence of the experimental technique on succes rate of the intervention, fluoroscopy time, radiation exposure, Major adverse cardiovascular event and tamponades (Safety) | 1 month
  Safety includes success of the intervention, fluoroscopy time, radiation exposure, Major adverse cardiovascular event and tamponades
Incidence of the experimental technique on direct and indirect costs (Cost-effectiveness) | 1 month
  Study costs includes direct costs (material used for the rapid pacing) and indirect costs (medical complications)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Faurie, Principal Investigator — Centre Recherche Cardio Vasculaire Alpes; Thierry Lefèvre, Principal Investigator — Massy
Locations (9):
- France (9):
  - CHU Clermont Ferrand, Clermont-Ferrand, Auvergne-Rhône-Alpes
  - Centre Hospitalier Annecy Genevois, Épagny, Auvergne-Rhône-Alpes
  - Clinique du Tonkin, Villeurbanne, Auvergne-Rhône-Alpes
  - Groupement Hospitalier Mutualiste de Grenoble, Grenoble, Isère
  - Hôpital privé Jacques Cartier, Paris, Massy
  - Clinique Saint-Hilaire, Rouen, Normandy
  - Clinique Pasteur, Toulouse, Occitanie
  - Institut Arnault Tzanck, Saint-Laurent-du-Var, Provence-Alpes-Côte d'Azur Region
  - Institut Mutualiste Montsouris, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adams DH, Popma JJ, Reardon MJ, Yakubov SJ, Coselli JS, Deeb GM, Gleason TG, Buchbinder M, Hermiller J Jr, Kleiman NS, Chetcuti S, Heiser J, Merhi W, Zorn G, Tadros P, Robinson N, Petrossian G, Hughes GC, Harrison JK, Conte J, Maini B, Mumtaz M, Chenoweth S, Oh JK; U.S. CoreValve Clinical Investigators. Transcatheter aortic-valve replacement with a self-expanding prosthesis. N Engl J Med. 2014 May 8;370(19):1790-8. doi: 10.1056/NEJMoa1400590. Epub 2014 Mar 29. PMID 24678937
- [Background] Arnold SV, Reynolds MR, Wang K, Magnuson EA, Baron SJ, Chinnakondepalli KM, Reardon MJ, Tadros PN, Zorn GL, Maini B, Mumtaz MA, Brown JM, Kipperman RM, Adams DH, Popma JJ, Cohen DJ; CoreValve US Pivotal Trial Investigators. Health Status After Transcatheter or Surgical Aortic Valve Replacement in Patients With Severe Aortic Stenosis at Increased Surgical Risk: Results From the CoreValve US Pivotal Trial. JACC Cardiovasc Interv. 2015 Aug 17;8(9):1207-1217. doi: 10.1016/j.jcin.2015.04.018. PMID 26292584
- [Background] Cribier A, Eltchaninoff H, Bash A, Borenstein N, Tron C, Bauer F, Derumeaux G, Anselme F, Laborde F, Leon MB. Percutaneous transcatheter implantation of an aortic valve prosthesis for calcific aortic stenosis: first human case description. Circulation. 2002 Dec 10;106(24):3006-8. doi: 10.1161/01.cir.0000047200.36165.b8. PMID 12473543
- [Background] Cribier A, Eltchaninoff H, Tron C, Bauer F, Agatiello C, Sebagh L, Bash A, Nusimovici D, Litzler PY, Bessou JP, Leon MB. Early experience with percutaneous transcatheter implantation of heart valve prosthesis for the treatment of end-stage inoperable patients with calcific aortic stenosis. J Am Coll Cardiol. 2004 Feb 18;43(4):698-703. doi: 10.1016/j.jacc.2003.11.026. PMID 14975485
- [Background] Eggebrecht H, Mehta RH, Kahlert P, Schymik G, Lefevre T, Lange R, Macaya C, Mandinov L, Wendler O, Thomas M. Emergent cardiac surgery during transcatheter aortic valve implantation (TAVI): insights from the Edwards SAPIEN Aortic Bioprosthesis European Outcome (SOURCE) registry. EuroIntervention. 2014 Dec;10(8):975-81. doi: 10.4244/EIJV10I8A165. PMID 24235321
- [Background] Faurie B, Abdellaoui M, Wautot F, Staat P, Champagnac D, Wintzer-Wehekind J, Vanzetto G, Bertrand B, Monsegu J. Rapid pacing using the left ventricular guidewire: Reviving an old technique to simplify BAV and TAVI procedures. Catheter Cardiovasc Interv. 2016 Nov 15;88(6):988-993. doi: 10.1002/ccd.26666. Epub 2016 Aug 11. PMID 27510946
- [Background] Gilard M, Eltchaninoff H, Iung B, Donzeau-Gouge P, Chevreul K, Fajadet J, Leprince P, Leguerrier A, Lievre M, Prat A, Teiger E, Lefevre T, Himbert D, Tchetche D, Carrie D, Albat B, Cribier A, Rioufol G, Sudre A, Blanchard D, Collet F, Dos Santos P, Meneveau N, Tirouvanziam A, Caussin C, Guyon P, Boschat J, Le Breton H, Collart F, Houel R, Delpine S, Souteyrand G, Favereau X, Ohlmann P, Doisy V, Grollier G, Gommeaux A, Claudel JP, Bourlon F, Bertrand B, Van Belle E, Laskar M; FRANCE 2 Investigators. Registry of transcatheter aortic-valve implantation in high-risk patients. N Engl J Med. 2012 May 3;366(18):1705-15. doi: 10.1056/NEJMoa1114705. PMID 22551129
- [Background] Karagoz T, Aypar E, Erdogan I, Sahin M, Ozer S, Celiker A. Congenital aortic stenosis: a novel technique for ventricular pacing during valvuloplasty. Catheter Cardiovasc Interv. 2008 Oct 1;72(4):527-30. doi: 10.1002/ccd.21695. PMID 18814234
- [Background] Lefevre T, Kappetein AP, Wolner E, Nataf P, Thomas M, Schachinger V, De Bruyne B, Eltchaninoff H, Thielmann M, Himbert D, Romano M, Serruys P, Wimmer-Greinecker G; PARTNER EU Investigator Group. One year follow-up of the multi-centre European PARTNER transcatheter heart valve study. Eur Heart J. 2011 Jan;32(2):148-57. doi: 10.1093/eurheartj/ehq427. Epub 2010 Nov 12. PMID 21075775
- [Background] Leon MB, Smith CR, Mack M, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Brown DL, Block PC, Guyton RA, Pichard AD, Bavaria JE, Herrmann HC, Douglas PS, Petersen JL, Akin JJ, Anderson WN, Wang D, Pocock S; PARTNER Trial Investigators. Transcatheter aortic-valve implantation for aortic stenosis in patients who cannot undergo surgery. N Engl J Med. 2010 Oct 21;363(17):1597-607. doi: 10.1056/NEJMoa1008232. Epub 2010 Sep 22. PMID 20961243
- [Background] Navarini S, Pfammatter JP, Meier B. Left ventricular guidewire pacing to simplify aortic balloon valvuloplasty. Catheter Cardiovasc Interv. 2009 Feb 15;73(3):426-7. doi: 10.1002/ccd.21810. No abstract available. PMID 19213097
- [Background] Popma JJ, Adams DH, Reardon MJ, Yakubov SJ, Kleiman NS, Heimansohn D, Hermiller J Jr, Hughes GC, Harrison JK, Coselli J, Diez J, Kafi A, Schreiber T, Gleason TG, Conte J, Buchbinder M, Deeb GM, Carabello B, Serruys PW, Chenoweth S, Oh JK; CoreValve United States Clinical Investigators. Transcatheter aortic valve replacement using a self-expanding bioprosthesis in patients with severe aortic stenosis at extreme risk for surgery. J Am Coll Cardiol. 2014 May 20;63(19):1972-81. doi: 10.1016/j.jacc.2014.02.556. Epub 2014 Mar 19. PMID 24657695
- [Background] Smith CR, Leon MB, Mack MJ, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Williams M, Dewey T, Kapadia S, Babaliaros V, Thourani VH, Corso P, Pichard AD, Bavaria JE, Herrmann HC, Akin JJ, Anderson WN, Wang D, Pocock SJ; PARTNER Trial Investigators. Transcatheter versus surgical aortic-valve replacement in high-risk patients. N Engl J Med. 2011 Jun 9;364(23):2187-98. doi: 10.1056/NEJMoa1103510. Epub 2011 Jun 5. PMID 21639811
- [Background] Thomas M, Schymik G, Walther T, Himbert D, Lefevre T, Treede H, Eggebrecht H, Rubino P, Colombo A, Lange R, Schwarz RR, Wendler O. One-year outcomes of cohort 1 in the Edwards SAPIEN Aortic Bioprosthesis European Outcome (SOURCE) registry: the European registry of transcatheter aortic valve implantation using the Edwards SAPIEN valve. Circulation. 2011 Jul 26;124(4):425-33. doi: 10.1161/CIRCULATIONAHA.110.001545. Epub 2011 Jul 11. PMID 21747054
- [Background] Walther T, Hamm CW, Schuler G, Berkowitsch A, Kotting J, Mangner N, Mudra H, Beckmann A, Cremer J, Welz A, Lange R, Kuck KH, Mohr FW, Mollmann H; GARY Executive Board. Perioperative Results and Complications in 15,964 Transcatheter Aortic Valve Replacements: Prospective Data From the GARY Registry. J Am Coll Cardiol. 2015 May 26;65(20):2173-80. doi: 10.1016/j.jacc.2015.03.034. Epub 2015 Mar 15. PMID 25787198
- [Background] Wenaweser P, Pilgrim T, Roth N, Kadner A, Stortecky S, Kalesan B, Meuli F, Bullesfeld L, Khattab AA, Huber C, Eberle B, Erdos G, Meier B, Juni P, Carrel T, Windecker S. Clinical outcome and predictors for adverse events after transcatheter aortic valve implantation with the use of different devices and access routes. Am Heart J. 2011 Jun;161(6):1114-24. doi: 10.1016/j.ahj.2011.01.025. Epub 2011 May 11. PMID 21641358
- [Background] Vogel R, Meier B. Emergent mechanical and electrical guidewire pacing of the right ventricle for aystole in the cardiac catheterization laboratory. J Invasive Cardiol. 2005 Sep;17(9):490. No abstract available. PMID 16145240
- [Derived] Faurie B, Souteyrand G, Staat P, Godin M, Caussin C, Van Belle E, Mangin L, Meyer P, Dumonteil N, Abdellaoui M, Monsegu J, Durand-Zaleski I, Lefevre T; EASY TAVI Investigators. Left Ventricular Rapid Pacing Via the Valve Delivery Guidewire in Transcatheter Aortic Valve Replacement. JACC Cardiovasc Interv. 2019 Dec 23;12(24):2449-2459. doi: 10.1016/j.jcin.2019.09.029. Epub 2019 Sep 28. PMID 31857014